CLINICAL TRIAL: NCT03337997
Title: A Pilot Study of Irreversible Electroporation for the Treatment of Upfront Resectable Pancreatic Cancer in the Head of the Pancreas
Brief Title: A Pilot Study of IRE for Resectable Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We have been unable to secure funding. Now we are in the middle of a pandemic.
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Michael Moser, Principal Investigator, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRE002
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Adenocarcinoma Resectable
Keywords: Irreversible Electroporation; Pancreatic Adenocarcinoma
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: Patients with biopsy-proven adenocarcinoma of the head of the pancreas deemed to be resectable by a multi-disciplinary team will be invited to participate.
Masking Description: CT scans and PET scans will be read by two radiologists and concensus obtained. The two radiologists will be unaware of prior chemo, patient age, original tumor size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): All patients in this pilot study are in the same group. All receive Irreversible Electroporation.
  Interventions: Procedure: Irreversible Electroporation

INTERVENTIONS:
Procedure: Irreversible Electroporation — Open Irreversible Electroporation by ultrasound guidance for tumors under 3 cm in diameter. Goal is to obtain an Amp rise of 12 or more
  Other Names: NanoKnife; IRE

SUMMARY:
The operation to remove certain pancreatic cancers (Whipple procedure), even in 2017, remains one of the most complicated surgeries done in the abdomen. It carries a 50% chance of a complication, even in the world's largest pancreatic surgery centres.

Saskatchewan is one of only two centres in Canada to have a promising new technology called Irreversible Electroporation (IRE) (NanoKnife®) available to our patients for the ablation (destruction) of cancers. IRE is different from other ablation treatments, including heat and even radiation, in that with IRE no heat is generated and there is minimal, if any, damage to nearby blood vessels, bowel, and ducts. Thus far, IRE has only been used as a "last resort" in cases where the pancreatic cancer cannot be removed with surgery, yet many patients whose tumor could likely be removed with a 'Whipple' have expressed a preference to undergo IRE instead of the Whipple procedure.

Our main research questions are: In comparison to Whipple procedure, is IRE an effective treatment of pancreatic cancer, and are complications reduced? Is IRE cost-effective? Based on the cases we have done and published series of IRE for stage III pancreatic cancer, we believe that IRE will be effective and safe in treating lesser stage (I and II) tumors in our proposed study.

This will be a pilot study of 12-15 patients, and all recruited patients will receive the IRE treatment and then be followed for up to 5 years for quality of life, recurrence, survival, and cost.

DETAILED DESCRIPTION:
* Subjects will receive a general anesthetic and will undergo a midline laparotomy and a careful inspection to ensure no distant metastases are obvious in the peritoneal cavity.
* Ultrasound-guided IRE of the pancreatic mass will be performed by interventional radiologist Dr. Chris Wall as per the protocol of Martin et al [ ].
* Subjects will be monitored for adverse events in the postoperative period until the time of discharge from the hospital, typically on the 5th or 6th day after the procedure.
* Adjuvant chemotherapy is recommended following the procedure but it is not mandatory.
* Patients will be assessed and offered single agent gemcitabine or combination of gemcitabine and capecitabine at the discretion of treating oncologists. It is recommended that patients begin treatment within 12 weeks after the procedure.
* Specific drug reductions and management of will be made in accordance with the published recommendations for gemcitabine or gemcitabine plus capecitabine.
* Patients will be scheduled for regular follow up and surveillance history and physical exam by the Hepatobiliary Surgeons Group.
* The same surveillance protocol that is used after the Whipple procedure will be followed: bloodwork at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months (complete blood count, electrolytes, creatinine, liver enzymes, Ca 19.9) and imaging (Chest Xray and CT abdomen at 3 months, followed by a PET scan at 6 months, CT scan at 9 and 12 months, then yearly CT or MRI).
* For study purposes, each scan will be re-reviewed by the same two radiologists with a goal of arriving at a consensus in each case.
* Two validated QOL questionnaires, the FACT-Hep, which is specific to hepatic and pancreatic diseases, and the more general FACT-G questionnaire will be administered preoperatively and at 3 and 12 months.
* Each IRE case will be matched 2:1 with patients undergoing the Whipple Procedure around the same time (within 12 months of each other) for non-locally advanced pancreatic cancer, matched by age +/- 5 years, gender, tumor size +/- 0.5 cm, and preoperative chemotherapy.
* Survival curves will be analyzed using the Kaplan-Meier method, and differences between groups will be assessed using log-rank test.
* Student's T test and the Mann-Whitney U test will be used for other comparisons between the two groups and p<0.05 will be taken to be significant. SPSS version 24 will be used for statistical analyses (SPSS Inc, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven pancreatic adenocarcinoma of the head of the pancreas.
* Age 18 to 75.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnancy
* Subjects who are medically unfit to receive a general anesthetic.
* Patients with cardiac arrhythmia other than rate controlled atrial fibrillation.
* Tumors greater than 3 cm.
* Unresectable or locally advanced pancreatic cancer.
* Patients with a high suspicion for lymph node metastasis or peripancreatic pathologic (> 1 cm) lymph nodes on imaging.
* Metastatic pancreatic carcinoma, including unexpected peritoneal or liver metastases discovered at the time of laparotomy for planned IRE.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years
  Disease Free Survival
Complications | 3 months
  recorded and classified

SECONDARY OUTCOMES:
Length of Stay | 1 month
  LOS
Quality of Life (Functional Assessment of Cancer Therapy- for Hepatobiliary and Pancreatic Cancers) questionnaire | preoperatively, 3 months, 12 months
  This is a validated measure of quality of life in patients who have hepato-pancreatico-biliary cancers, and includes 45 items that the patient scores on a scale of 0-4, with 4 being very symptomatic and 0 being asymptomatic. Higher scores imply a worse quality of life.
Time to recurrence | 5 years
  TTR
Overall Survival | 5 years
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided